CLINICAL TRIAL: NCT03094182
Title: Efficacy of Intravenous Iron Therapy in Maintaining Hemoglobin Concentration on Patients Undergoing Bimaxillary Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2016-1146
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Facial Asymmetry; Retrognathism; Prognathism
MeSH Terms: conditions — Facial Asymmetry; Retrognathia; Prognathism | interventions — iron isomaltoside 1000; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iron group (Experimental): Patients in the iron group are given Intravenous iron isomaltoside during operation.
  Interventions: Drug: Iron Isomaltoside 1000
- control group (Placebo Comparator): Patients in the control group receive the same volume of normal saline during operation.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — Randomly selected patients of the monofer group are given 1000mg of iron isomaltoside, which are mixed in 100ml normal saline, intravenous after induction for 30 minutes.
  Other Names: monofer®
  Arms: iron group
Drug: Normal saline — Randomly selected patients in the control group receive an equivalent volume of normal saline as a placebo.
  Arms: control group

SUMMARY:
The aim of this study is to evaluate the effect of Intravenous iron isomaltoside on maintaining hemoglobin concentration in patients undergoing bimaxillary orthognathic surgery. Fifty-eight patients, aged 19 to 40 years, scheduled for Bimaxillary orthognathic surgery will be divided into monofer (n=29) and control (n=29) groups. Randomly selected patients of the ulinastatin group are given intravenous iron isomaltoside. In contrast, patients in the control group receive an equivalent volume of normal saline as a placebo. The primary endpoints are postoperative hemoglobin concentration.

DETAILED DESCRIPTION:
Bimaxillary orthognathic surgery is widely used to correct dentofacial anomaly and bimaxillary prognathism. However, the complicated vascularity of the surgical site and limited visual field can lead to unexpected bleeding. Intravenous iron isomaltoside 1000 (monofer®) significantly increased the hemoglobin level and prevented anemia 4 weeks after cardiac surgery. The aim of this study is to evaluate the effect of Intravenous iron isomaltoside on maintaining hemoglobin concentration in patients undergoing bimaxillary orthognathic surgery. Fifty-eight patients, aged 19 to 40 years, scheduled for Bimaxillary orthognathic surgery will be divided into monofer (n=29) and control (n=29) groups. Randomly selected patients of the ulinastatin group are given intravenous iron isomaltoside. In contrast, patients in the control group receive an equivalent volume of normal saline as a placebo. The primary endpoints are postoperative hemoglobin concentration.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo bimaxillary orthognathic surgery
* American Society of Anesthesiologists (ASA) physical status I-II

Exclusion Criteria:

* hematologic disease
* renal-related anemia
* hepatitis
* pregnancy
* hypersensitivity to iron
* severe atopic disease
* allergic to drugs

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
postoperative hemoglobin level | 1 day after surgery
  Postoperative hemoglobin concentration
postoperative hemoglobin level | 2 weeks after surgery
  Postoperative hemoglobin concentration
postoperative hemoglobin level | 4 weeks after surgery
  Postoperative hemoglobin concentration

SECONDARY OUTCOMES:
hematogenous function | 1 day after surgery
  the hematogenous function measured by serum iron, ferritin, transferrin saturation, and total iron binding capacity, reticulocyte
hematogenous function | 2 weeks after surgery
  the hematogenous function measured by serum iron, ferritin, transferrin saturation, and total iron binding capacity, reticulocyte
hematogenous function | 4 weeks after surgery
  the hematogenous function measured by serum iron, ferritin, transferrin saturation, and total iron binding capacity, reticulocyte
quality of life(LASA) | 1 day after surgery
  The quality of life measured by LASA(Linear Analogue Self Assessment) questionnaire.
  LASA includes five simple items, each of which targets a specific domain of quality of life. Five single items(overall, physical, emotional, spiritual, intellectual) asking respondents to rate, on zero to ten scales, their perceived level of functioning.
quality of life(LASA) | 2 weeks after surgery
  The quality of life measured by LASA(Linear Analogue Self Assessment) questionnaire.
  LASA includes five simple items, each of which targets a specific domain of quality of life. Five single items(overall, physical, emotional, spiritual, intellectual) asking respondents to rate, on zero to ten scales, their perceived level of functioning.
quality of life(LASA) | 4 weeks after surgery
  The quality of life measured by LASA(Linear Analogue Self Assessment) questionnaire.
  LASA includes five simple items, each of which targets a specific domain of quality of life. Five single items(overall, physical, emotional, spiritual, intellectual) asking respondents to rate, on zero to ten scales, their perceived level of functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansson PI, Rasmussen AS, Thomsen LL. Intravenous iron isomaltoside 1000 (Monofer(R)) reduces postoperative anaemia in preoperatively non-anaemic patients undergoing elective or subacute coronary artery bypass graft, valve replacement or a combination thereof: a randomized double-blind placebo-controlled clinical trial (the PROTECT trial). Vox Sang. 2015 Oct;109(3):257-66. doi: 10.1111/vox.12278. Epub 2015 Apr 20. PMID 25900643
- [Background] Kalra PA, Bhandari S. Efficacy and safety of iron isomaltoside (Monofer((R))) in the management of patients with iron deficiency anemia. Int J Nephrol Renovasc Dis. 2016 Mar 10;9:53-64. doi: 10.2147/IJNRD.S89704. eCollection 2016. PMID 27022297
- [Background] Oh AY, Seo KS, Lee GE, Kim HJ. Effect of preoperative autologous blood donation on patients undergoing bimaxillary orthognathic surgery: a retrospective analysis. Int J Oral Maxillofac Surg. 2016 Apr;45(4):486-9. doi: 10.1016/j.ijom.2015.11.008. Epub 2015 Dec 8. PMID 26678802
- [Background] Litton E, Xiao J, Ho KM. Safety and efficacy of intravenous iron therapy in reducing requirement for allogeneic blood transfusion: systematic review and meta-analysis of randomised clinical trials. BMJ. 2013 Aug 15;347:f4822. doi: 10.1136/bmj.f4822. PMID 23950195
- [Background] Choi BK, Yang EJ, Oh KS, Lo LJ. Assessment of blood loss and need for transfusion during bimaxillary surgery with or without maxillary setback. J Oral Maxillofac Surg. 2013 Feb;71(2):358-65. doi: 10.1016/j.joms.2012.04.012. Epub 2012 Jun 16. PMID 22705218